CLINICAL TRIAL: NCT00402584
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled, Parallel Group Study to Examine the Efficacy and Safety of Meridia (Sibutramine Hydrochloride) in Binge-Eating Disorder
Brief Title: A Study to Examine the Efficacy and Safety of Meridia® (Sibutramine Hydrochloride) in Binge-Eating Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SB237
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Last update posted 2007-08-31 (Estimated); Status verified 2007-08

CONDITIONS: Binge Eating Disorder; Obesity
MeSH Terms: conditions — Binge-Eating Disorder; Obesity | interventions — sibutramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: sibutramine

SUMMARY:
The purpose of this study is to examine the safety and efficacy of sibutramine in preventing binge eating episodes. Additionally the study aim is to evaluate the safety and efficacy of sibutramine in reducing body weight in subjects with binge-eating disorder.

ELIGIBILITY:
Inclusion Criteria:

* Participants were men and women
* between the ages of 18 and 65
* with Body Mass Index (BMI) <45 kg/m2
* who met DSM-IV criteria for BED

Exclusion Criteria:

* Participants were excluded
* for blood pressure >140/90 mm Hg
* with pulse >95 beats/min
* history of stroke, narrow angle glaucoma, cardiac disease, seizures, renal or hepatic dysfunction
* use of insulin, medications known to affect body weight, or certain psychoactive medications (monoamine oxidase inhibitors, lithium, SSRIs, opioids)
* current participation in a weight loss program
* surgical treatment for obesity
* bulimia nervosa or purging in the past 6 months
* alcohol or drug abuse in the past 12 months
* current psychiatric condition being treated with a psychoactive agent
* current major depressive disorder
* history of anorexia nervosa, psychosis, bipolar disorder, or suicide attempts
* psychotherapy within the previous 2 months
* Women were excluded if they were pregnant, lactating, or if fertile, not practicing adequate contraceptive precautions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2000-08

PRIMARY OUTCOMES:
The frequency of binge eating episodes (binges/week), defined as the mean number of binges per week in 2-week intervals | 6 months

SECONDARY OUTCOMES:
Change from baseline in frequency of binge days (or mean days per week when the participant had one or more binges) | 6 months
Change from baseline in Body Weight | 6 months
Change from baseline in BMI | 6 months
Change from baseline in global improvement | 6 months
Change from baseline in eating pathology (TFEQ) | 6 months
Change from baseline in quality of life (IWQOL-Lite). | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bacher, MD, Study Director — Abbott

REFERENCES:
- [Derived] Wilfley DE, Crow SJ, Hudson JI, Mitchell JE, Berkowitz RI, Blakesley V, Walsh BT; Sibutramine Binge Eating Disorder Research Group. Efficacy of sibutramine for the treatment of binge eating disorder: a randomized multicenter placebo-controlled double-blind study. Am J Psychiatry. 2008 Jan;165(1):51-8. doi: 10.1176/appi.ajp.2007.06121970. Epub 2007 Dec 3. PMID 18056225